CLINICAL TRIAL: NCT04094649
Title: This is a Single-site, Double-blind, Randomized, Prospective, Sham-controlled, Crossover Early Feasibility Study to Determine Whether Ultrasound Vagus Nerve Stimulation (uVNS) Inhibits Postprandial Hyperglycemia in Humans
Brief Title: Acute Study of Effect of Ultrasound Vagus Nerve Stimulation on Glycemia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending funding
Sponsor: Aucta Technologies, Inc. (Industry)
Collaborators: STATKING Clinical Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: AT-C-19-01
Record Dates: First submitted 2019-08-06; First posted 2019-09-19 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a single-site, double-blind, randomized, prospective, sham-controlled, crossover early feasibility study to determine whether uVNS inhibits postprandial hyperglycemia in humans. Adults with DMT2 will be recruited and randomized to active uVNS or sham uVNS across two sessions according to a 2x2 crossover design.
Who Masked: Participant, Investigator
Masking Description: Randomization will be assigned by the clinical research facility. One of the two experimenters will be blinded. The unblinded experimenter is needed to aim the stimulation to the vagus nerve or sham location. The blinded experimenter will acquire, process, and analyze all data.
  Participants will be told that they may or may not feel the stimulation. The uVNS probe will be placed on their neck for each stimulation burst with the unblinded experimenter control-ling whether active or sham uVNS is delivered as determined by the crossover assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sham vs Active Stimulation Positions (Sham Comparator): Adults with Diabetes Mellitus Type 2 (DMT2) will be recruited and randomized to active uVNS or sham across two sessions according to a 2x2 crossover design. Sham uVNS will be delivered with the same stimulation parameters as active uVNS, but will be targeted to the left sternocleidomastoid muscle ~2 cm away from the vagus nerve.
  Interventions: Device: Ultrasound Vagus Nerve Stimulation (DECIMA)
- Active uVNS (Active Comparator): Active stimulations will be targeted with the ultrasound beam of the DECIMA device .Active uVNS will be delivered to the left cervical vagus nerve following the OGTT through the 60-min time point.
  Interventions: Device: Ultrasound Vagus Nerve Stimulation (DECIMA)

INTERVENTIONS:
Device: Ultrasound Vagus Nerve Stimulation (DECIMA) — This is a single-site, double-blind, randomized, prospective, sham-controlled, crossover early feasibility study to determine whether ultrasound Vagus Nerve Stimulation (uVNS) inhibits postprandial hyperglycemia in humans.

SUMMARY:
This is an early feasibility study to evaluate the proof of concept of modulation of glycemia by non-invasive ultrasound vagus nerve stimulation. This protocol is exploratory in nature, therefore it is not intended to capture statistically valid results or test statistical hypotheses. However, statistical analysis of the primary endpoint will be performed to allow more critical reflection of the data and to estimate the treatment effect for consider-ation in further studies.

DETAILED DESCRIPTION:
The DECIMA device comprises an array of two focused ultra-sound applicators arranged with overlapping foci to deliver acoustic energy to a known focal depth within tissue. The focused ultrasound applicators are each comprised of an ultra-sound-emitting piezoelectric element coupled to a focusing lens. The array of the DECIMA device is coupled with an ultra-sound imaging system to locate the cervical vagus nerve, and a control system to deliver short bursts of ultrasound energy that are controlled by the operator in time and intensity.

The imaging system and the array of applicators are calibrated together, so the power is focused at a known location relative to the imaging system screen. Each focused applicator's lens is joined to an ultrasound coupling cylinder filled with water. Each coupling cylinder is lined with thin plastic film at the skin. The ultrasound output power of the applicators is monitored by each applicator's control unit which includes a display of the ultrasound intensity.

To perform ultrasound stimulation, ultrasound gel is placed on the skin over the nerve area in the neck. Then the coupling cylinders and imaging transducer are placed against the gel, then the DECIMA position is fixed in place by a support arm.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any of the screening procedures
* Willingness to comply with all study procedures and available for the duration of the study
* Male or female age between 21 and 60 years old, inclusive
* Diabetes Mellitus Type 2 for at least 1 year

Exclusion Criteria:

* HbA1c greater than 10.5%
* Medical treatment regimen with insulin
* Medical treatment with antiinflammatory drugs such as Disease-Modifying Antirheumatic Drugs (DMARDs), i.e. Methotrexate and Cytokine-inhibitors, e.g. Adalimumab, and Etanercept.
* Clinically significant neuropathy in the opinion of the investigator or as documented in the subject's medical history
* Abundant fat tissue in neck, as evidenced by a neck circumference of more than 20''
* Clinically significant surgical procedure(s) or skin lesion(s) in neck that would affect subject safety or placement of device
* Prior vagotomy
* History of clinically significant vasovagal syncope or presyncope
* Use of electrically active implanted medical device
* History of heat stroke or any heat intolerance that is deemed clinically significant in the opinion of the investigator
* History of renal dysfunction or a glomerulonephropathy defined as either nephritic or nephrotic syndrome, including estimated glomerular filtration rate of <30 mL/min
* Clinically significant cardiovascular condition or problem that in the opinion of the investigator would interfere with the study data or affect patient safety (e.g. uncontrolled hypertension, congestive heart failure, or documented evidence of prior coronary artery disease).
* Pregnancy or plans to become pregnant while participating in the study, as determined by urine pregnancy test conducted at the screening visit for women of childbearing potential. A woman of childbearing potential is defined as a premenopausal female capable of becoming pregnant. This includes women on oral, injectable, or mechanical contraception; women who are single; women whose husbands have been vasectomized or whose husbands have received or are utilizing mechanical contraceptive devices.
* Uncontrolled asthma or obstructive lung disease.
* History of sepsis
* Significant cardiac rhythm disturbances in the opinion of the investigator based on an ECG.
* GI surgery that could have lacerated any branch of the vagus nerve, i.e. cholecystectomy, gastrectomy, pancreatic surgery, etc.
* Other conditions that could impair the patient's ability to participate in the study according to the investigator's opinion.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose Area Under the Curve (AUC, mg/dL ● hours) from baseline to 3 hours after an Oral Glucose Tolerance Test (OGTT) with Ultrasonic Vagus Nervous Stimulation (uVNS).hyperglycemia | Change from baseline in the 3-hour mean glucose AUC following an OGTT
  The DECIMA device comprises an array of two focused ultra-sound applicators arranged with overlapping foci to deliver acoustic energy to a known focal depth within tissue.

SECONDARY OUTCOMES:
Change in whole blood lipospolysaccharide-induced TNF-Alpha (pg/mL) production from base line to 4 hours post stimulation. | Change in mean Whole Blood Lipopolysaccharide-Induced TNF production from baseline to four (4) hours post-stimulation
  Inhibits postprandial hyperglycemia in patients with Diabetes Mellitus Type 2 via a temperature-medicated mechanism.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Tejada, MD, PI, Principal Investigator — Synexus
Locations (1):
- Cognitive Clinical Trials, LLC, Scottsdale, Arizona, United States